CLINICAL TRIAL: NCT02709304
Title: Exploring the Potential Efficacy of Lidocaine Gel in Reducing Discomfort in Patients Undergoing Surgical Procedures Requiring Foley Catheter Placement
Brief Title: Efficacy of Lidocaine Gel in Reducing Foley Catheter Discomfort in Surgical Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 693571
Record Dates: First submitted 2016-03-09; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Urinary Catheter Discomfort in Surgical Patients
Keywords: urinary catheter discomfort

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Gel (Placebo Comparator): Standard gel not containing local anesthetic used to insert urinary catheters.
  Interventions: Drug: standard gel
- Lidocaine Gel (Experimental): lidocaine containing gel uses to insert urinary catheters
  Interventions: Drug: Lidocaine gel

INTERVENTIONS:
Drug: Lidocaine gel — Gel used for insertion of urinary catheter containing local anesthetic to determine if patients have less discomfort postoperatively when this is used
  Other Names: Urojet
  Arms: Lidocaine Gel
Drug: standard gel — Standard gel that is used to insert a urinary catheter that does not contain local anesthetic
  Arms: Standard Gel

SUMMARY:
This study will evaluate whether lidocaine gel for urinary catheter insertion would decrease pain and discomfort associate with Foley catheters upon awakening from general anesthesia in the post anesthesia care unit. As a secondary objective, the study will evaluate bacterial colony counts from urine obtained from the surgical patients after insertion of the Foley catheter prior to prophylactic antimicrobial administration.

ELIGIBILITY:
Inclusion Criteria:

* Males requiring catheterization for surgical procedures scheduled for less than 4 hours.

Exclusion Criteria:

* Females, patients with preexisting urological conditions, and infections

Ages: 19 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Decrease postoperative urinary catheter related discomfort | Within 1 hour of emergence from general anesthetic
  Subject and objective pain scale

SECONDARY OUTCOMES:
decreased incidence of bacteriuria | immediate post catheter insertion and at 2 hour time point
  Urine culture and colony counts

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Reisbig, MD PhD, Principal Investigator — Creighton University School of Medicine / CHI Health

IPD SHARING:
Plan to Share IPD: Undecided